CLINICAL TRIAL: NCT05083845
Title: The Effect of Different Local Anesthetic Volumes for Thoracotomy Patients With Erector Spinae Plane Block
Brief Title: The Effect of Different Local Anesthetic Volumes on Postoperative Analgesia for Thoracotomy Patients With Erector Spinae Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Musa Zengin, Principal İnvestigator, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E.Kurul-E1-21-1964
Record Dates: First submitted 2021-10-04; First posted 2021-10-19 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Erector Spinae Plane Block; Local Anesthetic; Thoracotomy; Postoperative Analgesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block with 20 ml %0.25 Bupivacaine (Active Comparator): Following the visualization of the anatomical structures, the nerve block needle was advanced via the in-plane technique beneath the erector spinae muscles until the interfascial space was reached. After hydrodissection with 2 ml normal saline, 20 ml 0.25% bupivacaine was injected into the area.
  Interventions: Procedure: Same blocks with different local anesthetic volume
- Erector Spinae Plane Block with 30 ml %0.25 Bupivacaine (Active Comparator): Following the visualization of the anatomical structures, the nerve block needle was advanced via the in-plane technique beneath the erector spinae muscles until the interfascial space was reached. After hydrodissection with 2 ml normal saline, 30 ml 0.25% bupivacaine was injected into the area.
  Interventions: Procedure: Same blocks with different local anesthetic volume

INTERVENTIONS:
Procedure: Same blocks with different local anesthetic volume — Erector spinae plane block with different local anesthetic volumes will be applied to the patients under real-time ultrasound guidance.

SUMMARY:
It is widely accepted that thoracotomy causes severe acute pain. This increases the frequency of postoperative pulmonary complications and postoperative morbidity. Many analgesic methods have been proposed for thoracotomy pain, including thoracic epidural analgesia (TEA), thoracic paravertebral block (TPVB), intercostal nerve blocks (ICSB), erector spinae plane block (ESPB), serratus anterior plane block (SAPB). Among these methods, ultrasound-guided TPVB and ESPB are the most used methods. TPVB has left its place to newer techniques such as ESPB due to its proximity to the pleura and its deeper location. ESPB is more superficial, easy to access, and less likely to have complications. In addition, ESPB application is increasing in patients who underwent thoracotomy and VATS. There is no consensus on the dose of analgesia in these studies. There are studies on volumes between 10 ml and 40 ml in the literature. In this study, it was aimed to compare the volumes of 20 ml and 30 ml containing local anesthetic at the same concentration (0.25% bupivacaine) of ESPB block to be performed with USG in patients who underwent thoracotomy.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* ASA physical status I-II-III
* BMI 18 to 30 kg/m2
* Elective thoracotomy surgery

Exclusion Criteria:

* Patient refusing the procedure
* Emergency surgery
* History of chronic opioid or analgesic used

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-07-09 (Actual)

PRIMARY OUTCOMES:
Pain Scores | 48 hours after surgery
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at 1st, 2nd, 4th, 8th, 16th, 24th and 48th hours after surgery.

SECONDARY OUTCOMES:
Morphine Consumption | 24 hours after surgery
  Morphine consumption for 24 hours will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Atatürk Chest Disease and Chest Surgery Training and Research Hospital, Keçiören, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zengin M, Sazak H, Baldemir R, Ulger G, Arican D, Kaybal O, Alagoz A. Comparison of analgesic efficacy of different local anesthetic volumes for erector spinae plane block in thoracotomy patients; a prospective randomized trial. BMC Anesthesiol. 2023 Feb 6;23(1):42. doi: 10.1186/s12871-023-02004-4. PMID 36747119